CLINICAL TRIAL: NCT03863223
Title: A Phase 3,Randomized, Double-blinded, Placebo-controlled Study to Evaluate Efficacy and Safety of Pyrotinib Plus Trastuzumab and Docetaxel Versus Placebo Plus Trastuzumab and Docetaxel in Patients With HER2 Positive MBC.
Brief Title: A Study of Pyrotinib in Combination With Trastuzumab and Docetaxel in Patients With HER2 Metastatic Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-BLTN-III-MBC-C
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Trastuzumab; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- A (Experimental): Pyrotinib Plus trastuzumab and docetaxel
  Interventions: Drug: Pyrotinib, Trastuzumab, Docetaxel
- B (Placebo Comparator): Placebo plus trastuzumab and docetaxel
  Interventions: Drug: Placebo, Trastuzumab, Docetaxel

INTERVENTIONS:
Drug: Pyrotinib, Trastuzumab, Docetaxel — Pyrotinib 400mg orally daily until progressive disease
  Arms: A
Drug: Placebo, Trastuzumab, Docetaxel — Placebo 400mg orally daily until progressive disease
  Arms: B

SUMMARY:
This is a randomized, double-blinded, multicenter phase 3 clinical trial to evaluate the efficacy and safety of pyrotinib plus trastuzumab plus docetaxel versus placebo plus trastuzumab plus docetaxel in patients who have HER2 positive metastatic breast cancer and have not received systemic anticancer therapy for advanced disease.

ELIGIBILITY:
Inclusion Criteria:

1. HER2 positive recurrent or metastasis breast cancer.
2. Patients with measurable disease are eligible.
3. Eastern Cooperative Oncology Group(ECOG) performance status 0 or 1.
4. Adequate organ function.
5. Signed, written inform consent obtained prior to any study procedure.

Exclusion Criteria:

1. History of anti-cancer therapy for MBC（with the exception of one prior hormonal regimen for MBC）.
2. History of HER tyrosine kinase inhibitors or monoclonal antibody for breast cancer in any treatment setting，except trastuzumab used in the neo-adjuvant or adjuvant setting.
3. Assessed by the investigator to be unable receive systemic chemotherapy.
4. History of other malignancy within the last 5 years，except for carcinoma in situ of cervix，basal cell carcinoma or squamous cell carcinoma of the skin that has been previously treated with curative intent.
5. Pregnant or lactating women，or for women of childbearing potential unwilling to use a highly-effective contraception during of the study treatment and for at least 7 months after the last dose of study treatment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
PFS | Approximately 42 months
  Progression Free Survival

SECONDARY OUTCOMES:
AEs+SAEs | From the first drug administration to within 28 days for the last treatment
  Adverse Events and Serious Adverse Events
OS | Up to 2 years
  Overall Survival
ORR | Approximately 42 months
  Objective Response Rate
DoR | Approximately 42 months
  Duration of Objective Response
CBR | From the start of randomization to 6 months
  Clinical Benefit rate

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital,Chinese Academy of Medical Science, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma F, Yan M, Li W, Ouyang Q, Tong Z, Teng Y, Wang Y, Wang S, Geng C, Luo T, Zhong J, Zhang Q, Liu Q, Zeng X, Sun T, Mo Q, Liu H, Cheng Y, Cheng J, Wang X, Nie J, Yang J, Wu X, Wang X, Li H, Ye C, Dong F, Wu S, Zhu X, Xu B; PHILA Investigators. Pyrotinib versus placebo in combination with trastuzumab and docetaxel as first line treatment in patients with HER2 positive metastatic breast cancer (PHILA): randomised, double blind, multicentre, phase 3 trial. BMJ. 2023 Oct 31;383:e076065. doi: 10.1136/bmj-2023-076065. PMID 37907210